CLINICAL TRIAL: NCT04045873
Title: A Prospective, Multicenter, Randomized Clinical Trial of Hemodynamic Support With ECMO and IABP Versus IABP Alone, in Complex High-risk Patients Undergoing Elective PCI(PIONEER Trial)
Brief Title: PIONEER Trial:Hemodynamic Support With ECMO and IABP in Elective Complex High-risk PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Bethune International Peace Hospital (Other); Beijing Anzhen Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The General Hospital of Northern Theater Command (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192060-F-1
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease; Heart Failure
Keywords: Complex high-risk patients; Percutaneous coronary intervention; Extracorporeal membrane oxygenation; Intra-aortic balloon pump
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure | interventions — Extracorporeal Membrane Oxygenation; Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECMO plus IABP (Experimental)
  Interventions: Device: extracorporeal membrane oxygenation
- IABP (Experimental)
  Interventions: Device: extracorporeal membrane oxygenation

INTERVENTIONS:
Device: extracorporeal membrane oxygenation — The VA-ECMO procedure will be performed by femoral artery access, and the IABP will then be implanted in the contralateral femoral artery.
  Other Names: intra-aortic balloon pump

SUMMARY:
To determine whether hemodynamic support combining VA-ECMO with IABP could mitigate the rates of Major Adverse Cardiovascular and Cerebrovascular Events (MACCEs), compared with IABP support alone, in patients undergoing elective and high-risk PCI.

DETAILED DESCRIPTION:
Percutaneous Coronary Intervention (PCI) supported by mechanical circulatory device may be a viable alternative for these patients with complex coronary artery disease combined with multiple comorbidities and poor hemodynamics. Extracorporeal Membrane Oxygenation (ECMO) can direct blood flow out of the body, oxygenate it, and then return it, to either completely or partially replace the function of the heart and lungs, and potentially increase the likelihood of functional recovery. Limitations of ECMO include lack of direct LV unloading, and increased LV afterload with subsequent LV overload, which in turn can increase myocardial oxygen demand and therefore limit any cardioprotective benefits . Measures to concurrently decrease LV afterload during ECMO, such as use of an Intra-Aortic Balloon Pump (IABP), may in theory offset some of the disadvantages of ECMO. To date, ECMO has most commonly been used in patients suffering from cardiac arrest and cardiogenic shock . As far as we are aware, there exist very limited reported data from monocentric observational studies and individual case reports on the use of ECMO for elective, high-risk PCI in the literature . More importantly, no previous randomized studies to evaluate the safety and efficacy of a strategy combining VA-ECMO and IABP during high-risk PCI have been conducted to date. Most importantly, the strategy of combined VA-ECMO and IABP has never been investigated in any randomized trial that we could find.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 years to 85 years who meet any one of the following criteria

  1. Unprotected left main coronary artery disease with severe LV dysfunction (EF<35% or NYHA grade Ⅲ and Ⅳ).
  2. Unprotected left main coronary artery disease without severe LV dysfunction (LVEF>35% or NYHA Ⅰ and Ⅱ) must meet at least two of the complex procedure criteria (see Section II below).
  3. 3-vessel disease with severe LV dysfunction (EF<35% or NYHA grade Ⅲ and Ⅳ) must meet at least two of the complex procedure criteria (see Section II below).

Criteria Defining a Complex Procedure

1. Bifurcation requiring PCI in two branches (including PTCA or stenting).
2. Calcification requiring atherectomy.
3. Tortuosity requiring device assistance.
4. Difficult CTO（J-CTO score≥2）.

Exclusion Criteria:

1. Acute myocardial infarction within the previous 48 hours.
2. Pre-procedure cardiac arrest within 24 hours of enrollment requiring CPR.
3. Cardiogenic shock.
4. Complications of acute myocardial infarction (including ventricular septal defect, severe mitral regurgitation, and intractable ventricular arrhythmias).
5. Contraindications to IABP or ECMO use, including significant iliac or femoral arterial disease and more than mild aortic regurgitation as seen on echocardiography.
6. Bleeding diathesis or warfarin therapy with an international normalized ratio greater than 2.5.
7. Active internal bleeding (including menstruation) within the past month.
8. Recent ischemic stroke within the past month diagnosed by CT or MRI.
9. Previous hemorrhagic stroke diagnosed by CT or MRI.
10. Allergy to aspirin, clopidogrel, heparin, ticagrelor or glycoprotein IIb/ IIIa inhibitors; thrombocytopenia.
11. Pregnancy.
12. Current enrollment in any other study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy end point is the composite rate of MACCE at peri-procedure, in-hospital, or within a 30-day follow-up post-discharge. | 30 days
  The composite primary end point components include angiographic failure rates of PCI, all-cause death, myocardial infarction, stroke or transient ischemic attack, any repeat revascularization procedure, acute renal insufficiency, major vascular complications, severe intraprocedural hypotension requiring therapy, cardiopulmonary resuscitation, or ventricular tachycardia requiring cardioversion.

SECONDARY OUTCOMES:
The rate of complete revascularization | intra-procedure
intra-procedure hemodynamics | intra-procedure
vascular access site and access-related complications | intra-procedure
major or life-threatening or disabling bleeding | 30 days
stroke or transient ischemic attack | 30 days
acute kidney injury | 30 days
MACCE at 6 months | 6 months
MACCE at 1 year | 1 year
MACCE at 2 years | 2 years
MACCE at 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, PhD, Principal Investigator — Xijing Hospital; Chunguang Qiu, MD, PhD, Study Director — The First Affiliated Hospital of Zhengzhou University; Leisheng Ru, MD, PhD, Study Director — Bethune International Peace Hospital; Jinghua Liu, MD, PhD, Study Director — Beijing Anzhen Hospital; Bo Yu, MD, PhD, Study Director — The Second Affiliated Hospital of Harbin Medical University; Quanming Jing, MD, PhD, Study Director — The General Hospital of Northern Theater Command; Chengxiang Li, MD, PhD, Principal Investigator — Xijing Hospital